CLINICAL TRIAL: NCT00855192
Title: Antenatal Depression Group Research Project: The Effectiveness of Mindfulness-based Relaxation and Interpersonal Therapy to Relieve Anxiety and Depression Symptoms in Pregnant Women.
Brief Title: Antenatal Relaxation Group for Anxiety and Depression Management
Acronym: ARG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Saskatchewan (Other)
Collaborators: Royal University Hospital Foundation, Saskatoon, SK, Canada (Unknown)
Responsible Party: Angela Bowen, RN, PhD Assistant Professor, College of Nursing, College of Medicine, Department of Psychiatry, University of Saskatchewan
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Beh #07-10
Record Dates: First submitted 2009-03-02; First posted 2009-03-04 (Estimated); Last update posted 2010-03-18 (Estimated); Status verified 2009-03

CONDITIONS: Anxiety; Depression
Keywords: anxiety; depression; pregnancy; antenatal; prenatal; mindfulness-based therapy; interpersonal therapy; support groups
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- mindfulness-based therapy (Experimental): mindfulness-based meditation
  Interventions: Behavioral: mindful meditation
- interpersonal therapy (Experimental): psycho-educational
  Interventions: Behavioral: interpersonal therapy

INTERVENTIONS:
Behavioral: mindful meditation — interpersonal and psycho-educational
  Arms: mindfulness-based therapy
Behavioral: interpersonal therapy — psycho-educational
  Arms: interpersonal therapy

SUMMARY:
Approximately 20% of pregnant women experience depression. Untreated depression during pregnancy is linked to decreased prenatal care, difficulties in the pregnancy, poorer outcomes for the baby, and developmental, language, and behaviour problems in the older child.

While medication can often offer relief, pregnant women suffering with depression are often reluctant to take medications that may affect the unborn baby. There is little research about the effectiveness of other treatments such as support groups.

The investigators project will provide relaxation groups for pregnant women with anxiety and depression. The group will provide a chance to get support from other pregnant women. Two health care specialists will provide information about anxiety and depression. They will also teach the skills for women to manage their symptoms. Women will be asked to complete a few questionnaires to evaluate their symptoms before, during, and after they join the group. They will also be asked to evaluate how the group met their needs.

DETAILED DESCRIPTION:
Pregnant women between 15-28 weeks, who speak english are invited to join an 8 week group to relieve anxiety and depression.

We have collected sociodemographic data, as well as social support, life events.

Outcome measures are a decrease in anxiety and depression-as measured by the Edinburgh Postnatal Depression Scale, the Cambridge Worry Scale, and the STAI-Trait Scale.

ELIGIBILITY:
Inclusion Criteria:

* 15 to 28 weeks pregnant and English speaking

Exclusion Criteria:

* Non-English speaking

Ages: 16 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Depression as measured by Edinburgh Postnatal Depression Scale and anxiety as measured by the State-Trait Anxiety Inventory and the Cambridge Worry Scale | Participants will be asked to complete the questionnaires before the group commences, at 4 weeks, at the end of the group, and 6 weeks postpartum.

CONTACTS AND LOCATIONS:
Overall Officials: Angela N Bowen, PhD, Principal Investigator — University of Saskatchewan
Locations (2):
- Canada (2):
  - Saskatoon Community Village, Saskatoon, Saskatchewan
  - University of Saskatchewan Department of Psychiatry, Saskatoon, Saskatchewan